CLINICAL TRIAL: NCT00868582
Title: The National Oncologic PET Registry
Acronym: NOPR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: World Molecular Imaging Society (formerly Academy of Molecular Imaging) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NOPR
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cancer
Keywords: Patients with proven or suspected cancer referred for NaF-18 PET to identify bone metastasis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FDG-PET: F-18 fluorodeoxyglucose (FDG-PET)
  Interventions: Other: PET scanning in cancer
- NaF-18 PET: F-18 sodum-fluoride (NaF-18 PET)
  Interventions: Other: PET scanning in cancer

INTERVENTIONS:
Other: PET scanning in cancer — Collection of institutional practice PET imaging data
  Other Names: NOPR

SUMMARY:
The Centers for Medicare & Medicaid Services (CMS), as the Federal agency that administers the Medicare program, only pays for positron emission tomography (PET) scans in patients with cancer for certain reasons and for certain types of cancer. This study was developed to help CMS determine if they should pay for PET scans for additional reasons and additional types of cancer. In order to collect the information needed to decide which other types of cancer should be covered by Medicare, CMS will provide payment for the otherwise non-covered PET scans of patients who are properly registered with the National Oncologic PET Registry (NOPR). This information will then be analyzed to determine the effect PET scans had on the way physicians planned to treat their patients.

DETAILED DESCRIPTION:
The National Oncologic PET Registry (NOPR) was developed in response to the Centers for Medicare & Medicaid Services (CMS) proposal to expand coverage for positron emission tomography with F-18 fluorodeoxyglucose (FDG-PET) to include cancers and indications not presently eligible for Medicare reimbursement. Under this coverage with evidence development (CED) program, Medicare reimbursement for these cancers can be obtained if the patient's referring physician and the provider submit data to a clinical registry to assess the impact of PET on cancer patient management. The NOPR implemented this registry for CMS. The NOPR is sponsored by the World Molecular Imaging Society (formerly the Academy of Molecular Imaging), and managed by the American College of Radiology through the American College of Radiology Imaging Network.

The original goal of the National Oncologic PET Registry was to assess the effect of positron emission tomography with F-18 fluorodeoxyglucose (FDG-PET) on referring physicians' plans of intended patient management for those cancers and indications not currently eligible for reimbursement from CMS. Data were collected from the referring physician before and after the PET study. If complete and timely data are reported to the NOPR within 30 days of the PET scan, the PET facility and interpreting physician (nuclear physician/radiologist) are eligible for reimbursement by CMS. Based in part on data obtained from the NOPR, CMS expanded coverage for FDG-PET in patients with cancer on April 3, 2009 and further expanded coverage on June 11, 2013. Specifically, on June 11, 2013, CMS issued a final decision memorandum ending the prospective data collection requirements under CED for all oncologic indications for FDG-PET. Overall accrual to the FDG-PET registry was nearly 288,000 scans.

On February 26, 2010, CMS announced its decision to cover the use NaF-18 PET to identify bone metastasis. Under this new policy, the use of NaF-18 PET would be covered only under an approved (CED) program. The NOPR obtained CMS approval to develop a registry for NaF-18 as an amendment to the then-existing NOPR for FDG-PET. The NaF-18 PET registry component of NOPR was activated for accrual on February 7, 2011. Estimated total accrual to the NaF-PET registry is 45,000 cases.

As with the registry for FDG-PET, the goal of the NaF-18 PET registry component is to assess the impact of this imaging examination on referring physicians' plans of intended management of patients with known or suspected osseous metastatic disease. Data are collected from the referring physician before and after the PET study, as well as from the interpreting physician. If complete and timely data are reported to the NOPR within 30 days of the PET scan, the PET facility and interpreting physician (nuclear physician/radiologist) are eligible for reimbursement by CMS.

ELIGIBILITY:
Inclusion Criteria:

* All Medicare beneficiaries who are referred for NaF-18 PET to identify bone metastasis are eligible to be included in the NOPR.

Exclusion Criteria:

* NaF-18 PET for other (non-oncologic) indications.
* NaF-18 PET performed as part of a clinical trial approved by CMS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medicare beneficiaries who are referred for NaF-18 PET (the FDG-PET arm of NOPR has completed enrollment)
Sampling Method: Non-Probability Sample
Enrollment: 333000 (Estimated)
Dates: Start 2006-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of PET on referring physicians' plans of intended patient management of patients with cancer types eligible for inclusion in the National Oncologic PET Registry. | PET Scans as ordered by treating physician per CMS frequency guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Hillner, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- American College of Radiology Imaging Network, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Hillner BE, Siegel BA, Liu D, Shields AF, Gareen IF, Hanna L, Stine SH, Coleman RE. Impact of positron emission tomography/computed tomography and positron emission tomography (PET) alone on expected management of patients with cancer: initial results from the National Oncologic PET Registry. J Clin Oncol. 2008 May 1;26(13):2155-61. doi: 10.1200/JCO.2007.14.5631. Epub 2008 Mar 24. PMID 18362365
- [Result] Hillner BE, Siegel BA, Shields AF, Liu D, Gareen IF, Hunt E, Coleman RE. Relationship between cancer type and impact of PET and PET/CT on intended management: findings of the national oncologic PET registry. J Nucl Med. 2008 Dec;49(12):1928-35. doi: 10.2967/jnumed.108.056713. Epub 2008 Nov 7. PMID 18997054
- [Result] Hillner BE, Siegel BA, Shields AF, Liu D, Gareen IF, Hanna L, Stine SH, Coleman RE. The impact of positron emission tomography (PET) on expected management during cancer treatment: findings of the National Oncologic PET Registry. Cancer. 2009 Jan 15;115(2):410-8. doi: 10.1002/cncr.24000. PMID 19016303
- [Result] Hillner BE, Siegel BA, Shields AF, Duan F, Gareen IF, Hanna L, Coleman RE. Impact of dedicated brain PET on intended patient management in participants of the national oncologic PET Registry. Mol Imaging Biol. 2011 Feb;13(1):161-5. doi: 10.1007/s11307-010-0427-5. PMID 21080232
- [Result] Hillner BE, Siegel BA, Hanna L, Shields AF, Duan F, Gareen IF, Quinn B, Coleman RE. Impact of 18F-FDG PET used after initial treatment of cancer: comparison of the National Oncologic PET Registry 2006 and 2009 cohorts. J Nucl Med. 2012 May;53(5):831-7. doi: 10.2967/jnumed.112.103911. Epub 2012 Mar 23. PMID 22448033
- [Result] Hillner BE, Tosteson TD, Tosteson AN, Wang Q, Song Y, Onega T, Hanna LG, Siegel BA. Intended versus inferred management after PET for cancer restaging: analysis of Medicare claims linked to a coverage with evidence development registry. Med Care. 2013 Apr;51(4):361-7. doi: 10.1097/MLR.0b013e318287d860. PMID 23481033
- [Result] Hillner BE, Tosteson AN, Tosteson TD, Wang Q, Song Y, Hanna LG, Siegel BA. Intended versus inferred care after PET performed for initial staging in the National Oncologic PET Registry. J Nucl Med. 2013 Dec;54(12):2024-31. doi: 10.2967/jnumed.113.123430. Epub 2013 Nov 12. PMID 24221994
- [Result] Hillner BE, Siegel BA, Hanna L, Duan F, Shields AF, Coleman RE. Impact of 18F-fluoride PET in patients with known prostate cancer: initial results from the National Oncologic PET Registry. J Nucl Med. 2014 Apr;55(4):574-81. doi: 10.2967/jnumed.113.130005. Epub 2014 Feb 27. PMID 24578240
- [Result] Hillner BE, Siegel BA, Hanna L, Duan F, Shields AF, Quinn B, Coleman RE. Impact of (18)F-Fluoride PET on Intended Management of Patients with Cancers Other Than Prostate Cancer: Results from the National Oncologic PET Registry. J Nucl Med. 2014 Jul;55(7):1054-61. doi: 10.2967/jnumed.113.135475. Epub 2014 May 12. PMID 24819422
- [Result] Hillner BE, Siegel BA, Hanna L, Duan F, Quinn B, Shields AF. 18F-fluoride PET used for treatment monitoring of systemic cancer therapy: results from the National Oncologic PET Registry. J Nucl Med. 2015 Feb;56(2):222-8. doi: 10.2967/jnumed.114.150391. Epub 2015 Jan 15. PMID 25593113